CLINICAL TRIAL: NCT00125034
Title: Open, Randomized, Controlled, Multicenter Phase II Study Comparing 5-FU/FA Plus Oxaliplatin (FOLFOX-4) Plus Cetuximab Versus 5-FU/FA Plus Oxaliplatin (FOLFOX-4) as First-line Treatment for Epidermal Growth Factor Receptor-expressing Metastatic Colorectal Cancer
Brief Title: Oxaliplatin and Cetuximab in First-line Treatment of Metastatic Colorectal Cancer (mCRC)
Acronym: OPUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62202-047
Record Dates: First submitted 2005-07-28; First posted 2005-07-29 (Estimated); Results first posted 2011-10-04 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2011-08

CONDITIONS: Neoplasm Metastasis; Colorectal Cancer
Keywords: FOLFOX-4; Cetuximab; First-line mCRC; EGFR positive; metastatic CRC
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms | interventions — Cetuximab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cetuximab Plus FOLFOX-4 (Experimental)
  Interventions: Biological: Cetuximab
- FOLFOX-4 Alone (Active Comparator)
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Biological: Cetuximab — Cetuximab will always be administered first, followed by oxaliplatin at least 1 hour later. Following completion of the oxaliplatin infusion or simultaneously with oxaliplatin folinic acid (FA) will be administered (at a dose of 200 mg/m^2, infused over 120 minutes, on day 1 and day 2, every two weeks) and then 5-Fluorouracil (5-FU) (as a bolus of 400 mg/m^2/day intravenously (IV) over 2-4 minutes followed by 600 mg/m^2/day infused over 22-hour, on day 1 and day 2, every two weeks).
  Until progression or unacceptable toxicity develops
  Arms: Cetuximab Plus FOLFOX-4
Drug: Oxaliplatin — Oxaliplatin will always be administered first or simultaneously with FA (at a dose of 200 mg/m^2, infused over 120 minutes, on day 1 and day 2, every two weeks) and then 5-FU (as a bolus of 400 mg/m^2/day IV over 2-4 minutes followed by 600 mg/m^2/day infused over 22-hour, on day 1 and day 2, every two weeks).
  Until progression or unacceptable toxicity develops
  Arms: FOLFOX-4 Alone

SUMMARY:
This is an open label, randomized, controlled, multicenter phase II study comparing 5-FU/FA + oxaliplatin (FOLFOX-4) + cetuximab versus 5-FU/FA + oxaliplatin as first-line treatment for epidermal growth factor receptor (EGFR)-expressing mCRC.

ELIGIBILITY:
Inclusion Criteria:

* First-line mCRC
* EGFR positive
* Bi-dimensional measurable index lesion

Exclusion Criteria:

* Previous exposure to EGFR-targeting therapy
* Previous oxaliplatin-based therapy
* Previous chemotherapy for colorectal cancer except adjuvant treatment with progression of disease documented > 6 months after end of adjuvant treatment
* Radiotherapy
* Surgery
* Any other investigational drug in the 30 days before randomization
* Brain metastasis and/or leptomeningeal disease
* Acute or sub-acute intestinal occlusion or history of inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2005-07; Primary Completion 2007-03 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bokemeyer, Prof. Dr., Principal Investigator — Klinik für Onkologie, Hämatologie und Knochenmarktransplantationen Universitätsklinikum Hamburg-Eppendorf, Germany
Locations (78):
- Austria (5):
  - Research Site, Graz
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Zams
- Belgium (8):
  - Research Site, Antwerp
  - Research Site, Bonheiden
  - Research Site, Bruges
  - Research Site, Hasselt
  - Research Site, Leuven
  - Research Site, Roeselare
  - Research Site, Turnhout
  - Research Site, ZU Gent
- France (7):
  - Research Site, Besançon
  - Research Site, Clermond Ferrand
  - Research Site, Clichy
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Rouen
  - Research Site, Strasbourg
- Germany (9):
  - Research Site, Aschaffenburg
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Hamburg
  - Research Site, Kiel
  - Research Site, Magdeburg
  - Research Site, Mannheim
  - Research Site, Nuremberg
  - Research Site, Tübingen
- Greece (3):
  - Research Site, Athens
  - Research Site, Loannina
  - Research Site, Thessaloniki
- Israel (6):
  - Research Site, Haifa
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Rehovot
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Italy (6):
  - Research Site, Brescia
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Pavia
  - Research Site, Rome
  - Research Site, Torino
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Opole
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Warsaw
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Santa Maira Da Feira
- Romania (5):
  - Research Site, Alba Iulia
  - Research Site, Bucurest
  - Research Site, Onești
  - Research Site, Oradea
  - Research Site, Timișoara
- Russia (6):
  - Research Site, Kazan'
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Obninsk
  - Research Site, Saint Petersburg
  - Research Site, Samara
- Spain (8):
  - Research Site, Bilbao
  - Research Site, Burgos
  - Research Site, Girona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Ourense
  - Research Site, Reus
  - Research Site, Valencia
- Ukraine (6):
  - Research Site, Dnipro
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Lviv
  - Research Site, Simferopol
  - Research Site, Vinnitsa

REFERENCES:
- [Result] Bokemeyer C, Bondarenko I, Makhson A, Hartmann JT, Aparicio J, de Braud F, Donea S, Ludwig H, Schuch G, Stroh C, Loos AH, Zubel A, Koralewski P. Fluorouracil, leucovorin, and oxaliplatin with and without cetuximab in the first-line treatment of metastatic colorectal cancer. J Clin Oncol. 2009 Feb 10;27(5):663-71. doi: 10.1200/JCO.2008.20.8397. Epub 2008 Dec 29. PMID 19114683
- [Result] Bokemeyer C, Bondarenko I, Hartmann JT, de Braud F, Schuch G, Zubel A, Celik I, Schlichting M, Koralewski P. Efficacy according to biomarker status of cetuximab plus FOLFOX-4 as first-line treatment for metastatic colorectal cancer: the OPUS study. Ann Oncol. 2011 Jul;22(7):1535-1546. doi: 10.1093/annonc/mdq632. Epub 2011 Jan 12. PMID 21228335

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First & last subject randomized: 27 Jul 2005 & 8 Mar 2006, respectively. Primary outcome and disease control rate cut-off dates 4 Aug 2006, others: 1 Mar 2007; except overall survival, KRAS overall survival and KRAS progression-free survival outcomes, metastatic surgery outcome and adverse events: 30 Nov 2008.
Pre-assignment Details: 629 subjects were prescreened, of whom 344 subjects were randomised. 338 subjects (Safety Population) received treatment. One subject was erroneously randomized, and was excluded from the ITT population (337 subjects).
Groups:
- Cetuximab Plus FOLFOX-4: Cetuximab plus 5-Fluorouracil(5-FU)/Folinic acid (FA) and oxaliplatin. Cetuximab will always be administered first, followed by oxaliplatin at least 1 hour later. Following completion of the oxaliplatin infusion or simultaneously with oxaliplatin FA will be administered (at a dose of 200 mg/m^2, infused over 120 minutes, on day 1 and day 2, every two weeks) and then 5-FU (as a bolus of 400 mg/m^2/day intravenously (IV) over 2-4 minutes followed by 600 mg/m^2/day infused over 22-hour, on day 1 and day 2, every two weeks). Until progression or unacceptable toxicity develops. Safety population: includes all treated subjects.
- FOLFOX-4 Alone: 5-FU/FA and oxaliplatin. Oxaliplatin will always be administered first or simultaneously with FA (at a dose of 200 mg/m^2, infused over 120 minutes, on day 1 and day 2, every two weeks) and then 5-FU (as a bolus of 400 mg/m^2/day IV over 2-4 minutes followed by 600 mg/m^2/day infused over 22-hour, on day 1 and day 2, every two weeks). Until progression or unacceptable toxicity develops. Safety population: includes all treated subjects.
Period: Overall Study
Arm/Group | Cetuximab Plus FOLFOX-4 | FOLFOX-4 Alone
Started | 170 (Randomized & treated. 1 subject was not randomized correctly and was excluded in the ITT population.) | 168 (Randomized & treated)
Completed | 170 | 168
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab Plus FOLFOX-4 | FOLFOX-4 Alone | Total
Number analyzed (Participants) | 169 | 168 | 337
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 96 | 109 | 205
  >=65 years | 73 | 59 | 132
Age, Continuous [Median (Full Range); unit: years] | 62.0 [24 to 82] | 60.0 [30 to 82] | 61.0 [24 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 76 | 156
  Male | 89 | 92 | 181
Region of Enrollment [Number; unit: participants] — Figures refer to randomized and treated participants
  participants
    Portugal | 0 | 3 | 3
    Spain | 19 | 16 | 35
    Ukraine | 24 | 25 | 49
    Austria | 16 | 9 | 25
    Russian Federation | 25 | 24 | 49
    Israel | 0 | 1 | 1
    Italy | 8 | 6 | 14
    France | 3 | 12 | 15
    Belgium | 12 | 6 | 18
    Poland | 30 | 31 | 61
    Romania | 18 | 13 | 31
    Germany | 14 | 22 | 36

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate - Independent Review Committee (IRC)
Description: The best overall response rate is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response as the best overall response according to radiological assessments (based on modified World Health Organisation (WHO) criteria) as assessed by an IRC.
Time Frame: Evaluations were performed every 6 weeks until progression, reported between day of first patient randomised, 27 Jul 2005, until cut-off date 4 August 2006
Population: Primary analysis on the Intent to Treat (ITT) population i.e. all randomized subjects who have received at least one dose of randomized treatment (allocation to treatment groups as randomized).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab Plus FOLFOX-4 | FOLFOX-4 Alone
Number analyzed (Participants) | 169 | 168
percentage of participants | 45.6 [37.9 to 53.4] | 35.7 [28.5 to 43.5]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFOX-4 vs FOLFOX-4 Alone; Assuming a difference in rate of best confirmed response of at least 20% between the 2 treatments, ie an approximately 70% response rate under cetuximab plus FOLFOX-4 & 50% under FOLFOX-4 alone for the stratum with ECOG PS0-1 & 66% and 45% respectively for the ECOG PS2 stratum, the common OddsR over the strata was expected to be 2.33. A sample size of approximately 146/group was calculated as necessary to detect a significant overall response of at least 2.33 at level α=0.05 with a power of 90%; Test type: Superiority or Other; p = 0.064, stratified Cochran-Mantel-Haenszel test; Stratified odds ratio and Cochran-Mantel-Haenszel (CMH) statistics were calculated considering the randomization strata; Odds Ratio (OR) = 1.516, 95% CI 2-sided [0.975 to 2.335]

2. Secondary Outcome: Best Overall Response Rate (Chinese V-Ki-ras2 Kirsten Rat Sarcoma Viral Oncogene Homolog (KRAS) Wild-Type Population)
Description: The best overall response rate is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response as the best overall response according to radiological assessments (based on modified WHO criteria) as assessed by an IRC.
Time Frame: Evaluations were performed every 6 weeks until progression, reported between day of first patient randomised, 27 Jul 2005, until cut-off date 1 Mar 2007
Population: KRAS Wild-Type population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab Plus FOLFOX-4 | FOLFOX-4 Alone
Number analyzed (Participants) | 82 | 97
percentage of participants | 57.3 [45.9 to 68.2] | 34.0 [24.7 to 44.3]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFOX-4 vs FOLFOX-4 Alone; Test type: Superiority or Other; p = 0.0027, stratified Cochran-Mantel-Haenszel test; Stratified odds ratio and Cochran-Mantel-Haenszel (CMH) statistics were calculated considering the randomization strata; Odds Ratio (OR) = 2.551, 95% CI 2-sided [1.380 to 4.717]

3. Secondary Outcome: Best Overall Response Rate (KRAS Mutant Population)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: KRAS Mutant population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab Plus FOLFOX-4 | FOLFOX-4 Alone
Number analyzed (Participants) | 77 | 59
percentage of participants | 33.8 [23.4 to 45.5] | 52.5 [39.1 to 65.7]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFOX-4 vs FOLFOX-4 Alone; Test type: Superiority or Other; p = 0.0290, stratified Cochran-Mantel-Haenszel test; Stratified odds ratio and Cochran-Mantel-Haenszel (CMH) statistics were calculated considering the randomization strata; Odds Ratio (OR) = 0.459, 95% CI 2-sided [0.228 to 0.924]

4. Secondary Outcome: Progression-free Survival Time
Description: Duration from randomization until radiological progression as assessed by an IRC (based on modified WHO criteria) or death due to any cause.
  Only deaths within 60 days of last tumor assessment are considered. Patients without event are censored on the date of last tumor assessment.
Time Frame: Time from randomisation to disease progression, death or last tumour assessment, reported between day of first patient randomised, 27 Jul 2005, until cut-off date 01 Mar 2007
Population: Primary analysis on ITT population i.e. all randomized subjects who have received at least one dose of randomized treatment (allocation to treatment groups as randomized).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus FOLFOX-4 | FOLFOX-4 Alone
Number analyzed (Participants) | 169 | 168
months | 7.2 [5.6 to 7.7] | 7.2 [6.0 to 7.8]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFOX-4 vs FOLFOX-4 Alone; Test type: Superiority or Other; p = 0.6170, Stratified Log Rank; Kaplan-Meier method used to estimate median OS time. HR was calculated using Cox proportional hazards model stratified by randomization strata; Hazard Ratio (HR) = 0.931, 95% CI 2-sided [0.705 to 1.230]

5. Secondary Outcome: Progression-free Survival Time (KRAS Wild-Type Population)
Description: as for outcome 4
Time Frame: Time from randomisation to disease progression, death or last tumour assessment, reported between day of first patient randomised, 27 Jul 2005, until cut-off date 30 Nov 2008
Population: KRAS Wild-Type population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus FOLFOX-4 | FOLFOX-4 Alone
Number analyzed (Participants) | 82 | 97
months | 8.3 [7.2 to 12.0] | 7.2 [5.6 to 7.4]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFOX-4 vs FOLFOX-4 Alone; Test type: Superiority or Other; p = 0.0064, Stratified Log Rank; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.567, 95% CI 2-sided [0.375 to 0.856]

6. Secondary Outcome: Progression-free Survival Time (KRAS Mutant Population)
Description: as for outcome 4
Time Frame: as for outcome 5
Population: KRAS Mutant population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus FOLFOX-4 | FOLFOX-4 Alone
Number analyzed (Participants) | 77 | 59
months | 5.5 [4.0 to 7.3] | 8.6 [6.5 to 9.4]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFOX-4 vs FOLFOX-4 Alone; Test type: Superiority or Other; p = 0.0153, Stratified Log Rank; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.720, 95% CI 2-sided [1.104 to 2.679]

7. Secondary Outcome: Overall Survival Time
Description: Time from randomization to death. Patients without event are censored at the last date known to be alive or at the clinical cut-off date, whatever is earlier.
Time Frame: Time from randomisation to death or last day known to be alive, reported between day of first patient randomised, 27 Jul 2005, until cut-off date 30 Nov 2008
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus FOLFOX-4 | FOLFOX-4 Alone
Number analyzed (Participants) | 169 | 168
months | 18.3 [14.8 to 20.4] | 18.0 [16.7 to 21.8]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFOX-4 vs FOLFOX-4 Alone; Test type: Superiority or Other; p = 0.9050, Stratified log rank; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.015, 95% CI 2-sided [0.791 to 1.303]

8. Secondary Outcome: Overall Survival Time (KRAS Wild-Type Population)
Description: as for outcome 7
Time Frame: Time from randomisation to death or last day known to be alive, reported between day of first patient randomised, 27 Jul 2005, until cut-off date 30 November 2008
Population: KRAS Wild-Type population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus FOLFOX-4 | FOLFOX-4 Alone
Number analyzed (Participants) | 82 | 97
months | 22.8 [19.3 to 25.9] | 18.5 [16.4 to 22.6]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFOX-4 vs FOLFOX-4 Alone; Test type: Superiority or Other; p = 0.3854, Stratified log rank; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.855, 95% CI 2-sided [0.599 to 1.219]

9. Secondary Outcome: Overall Survival Time (KRAS Mutant Population)
Description: as for outcome 7
Time Frame: as for outcome 8
Population: KRAS Mutant population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus FOLFOX-4 | FOLFOX-4 Alone
Number analyzed (Participants) | 77 | 59
months | 13.4 [10.5 to 17.7] | 17.5 [14.7 to 24.8]
Statistical Analysis 1: Comparison: Cetuximab Plus FOLFOX-4 vs FOLFOX-4 Alone; Test type: Superiority or Other; p = 0.2004, Stratified log rank; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.290, 95% CI 2-sided [0.873 to 1.906]

10. Secondary Outcome: Participants With No Residual Tumor After Metastatic Surgery
Description: No residual tumor after on-study surgery for metastases.
Time Frame: Time from first dose up to 30 days after the last dose of study treatment, reported between day of first patient randomised, 27 Jul 2005, until cut-off date 30 November 2008
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Cetuximab Plus FOLFOX-4 | FOLFOX-4 Alone
Number analyzed (Participants) | 169 | 168
participants | 8 | 4

11. Secondary Outcome: Disease Control Rate (Cut Off Date 4 August 2006)
Description: The disease control rate is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response + Stable Disease as best overall response according to radiological assessments as assessed by IRC (based on modified WHO criteria).
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab Plus FOLFOX-4 | FOLFOX-4 Alone
Number analyzed (Participants) | 169 | 168
percentage of participants | 85.2 [78.9 to 90.2] | 81.0 [74.2 to 86.6]

12. Secondary Outcome: Duration of Response
Description: Time from first assessment of Complete Response or Partial Response to disease progression or death (within 60 days of last tumor assessment).
  Patients without event are censored on the date of last tumor assessment. Tumor assessments based on modified WHO criteria.
Time Frame: Time from first assessment of Complete Response or Partial Response to disease progression,death or last tumor assessment, reported between day of first patient randomised, 27 Jul 2005, until cut-off date 01 Mar 2007
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus FOLFOX-4 | FOLFOX-4 Alone
Number analyzed (Participants) | 169 | 168
months | 9.0 [5.9 to 11.1] | 5.7 [5.4 to 7.7]

13. Secondary Outcome: Safety - Number of Patients Experiencing Any Adverse Event
Description: Please refer to Adverse Events section for further details
Time Frame: time from first dose up to 30 after last dose of study treatment, reported between day of first patient dose of study treatment, 27 Jul 2005, until cut-off date 30 Nov 2008
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Cetuximab Plus FOLFOX-4 | FOLFOX-4 Alone
Number analyzed (Participants) | 170 | 168
participants | 170 | 165

ADVERSE EVENTS:
Time Frame: Time from first dose up to 30 days after the last dose of study treatment.
Description: Treatment-emergent adverse events were defined as those with onset occurring at or after the first dosing day of study medication and up to 30 days after the last administration of any study drug or the clinical cut-off date.
Arm/Group | Cetuximab Plus FOLFOX-4 | FOLFOX-4 Alone
Serious Adverse Events (participants affected / at risk) | 61/170 | 43/168
Other Adverse Events (participants affected / at risk) | 170/170 | 165/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus FOLFOX-4 (N=170) | FOLFOX-4 Alone (N=168)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 0 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 4 | 3
LEUKOPENIA (Blood and lymphatic system disorders) | 3 | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 4 | 5
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 2 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 2 | 0
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 0
CONJUNCTIVITIS (Eye disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 1
ASCITES (Gastrointestinal disorders) | 2 | 0
COLITIS (Gastrointestinal disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 2 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 2
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 1
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 1
ILEUS (Gastrointestinal disorders) | 4 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 | 0
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 1 | 0
PERITONITIS (Gastrointestinal disorders) | 0 | 1
RECTAL STENOSIS (Gastrointestinal disorders) | 0 | 1
SUBILEUS (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 2 | 4
ASTHENIA (General disorders) | 3 | 1
CHEST PAIN (General disorders) | 1 | 0
FATIGUE (General disorders) | 1 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 1
INJECTION SITE REACTION (General disorders) | 1 | 0
MASS (General disorders) | 1 | 0
MUCOSAL INFLAMMATION (General disorders) | 1 | 0
OBSTRUCTION (General disorders) | 0 | 1
PYREXIA (General disorders) | 4 | 4
BILE DUCT STONE (Hepatobiliary disorders) | 0 | 1
CHOLANGITIS (Hepatobiliary disorders) | 1 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0
HEPATORENAL SYNDROME (Hepatobiliary disorders) | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 2 | 0
JAUNDICE (Hepatobiliary disorders) | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 5 | 2
ABSCESS NECK (Infections and infestations) | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 1
CATHETER RELATED INFECTION (Infections and infestations) | 0 | 1
CENTRAL LINE INFECTION (Infections and infestations) | 0 | 1
ERYSIPELAS (Infections and infestations) | 2 | 0
FEBRILE INFECTION (Infections and infestations) | 1 | 0
INFECTION (Infections and infestations) | 2 | 1
KIDNEY INFECTION (Infections and infestations) | 0 | 1
LUNG ABSCESS (Infections and infestations) | 1 | 0
PERITONITIS BACTERIAL (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 3 | 3
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 | 1
SEPSIS (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 | 0
TUBERCULOSIS (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 1 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 | 0
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 | 0
ANOREXIA (Metabolism and nutrition disorders) | 3 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 1
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 2 | 0
DIZZINESS (Nervous system disorders) | 0 | 1
EPILEPSY (Nervous system disorders) | 0 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 1 | 0
ALCOHOLIC PSYCHOSIS (Psychiatric disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
MEDIASTINAL HAEMATOMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 5 | 2
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ILEOCOLOSTOMY (Surgical and medical procedures) | 0 | 1
AXILLARY VEIN THROMBOSIS (Vascular disorders) | 1 | 0
CIRCULATORY COLLAPSE (Vascular disorders) | 0 | 1
EMBOLISM (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 2 | 0
HYPOTENSION (Vascular disorders) | 1 | 0
INTERMITTENT CLAUDICATION (Vascular disorders) | 1 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 0
THROMBOPHLEBITIS (Vascular disorders) | 0 | 1
VENOUS THROMBOSIS (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus FOLFOX-4 (N=170) | FOLFOX-4 Alone (N=168)
ANAEMIA (Blood and lymphatic system disorders) | 44 | 41
LEUKOPENIA (Blood and lymphatic system disorders) | 49 | 43
NEUTROPENIA (Blood and lymphatic system disorders) | 77 | 84
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 45 | 69
VERTIGO (Ear and labyrinth disorders) | 9 | 7
CONJUNCTIVITIS (Eye disorders) | 23 | 8
ABDOMINAL PAIN (Gastrointestinal disorders) | 30 | 29
CONSTIPATION (Gastrointestinal disorders) | 32 | 16
DIARRHOEA (Gastrointestinal disorders) | 81 | 68
DYSPEPSIA (Gastrointestinal disorders) | 9 | 9
NAUSEA (Gastrointestinal disorders) | 69 | 65
STOMATITIS (Gastrointestinal disorders) | 33 | 19
VOMITING (Gastrointestinal disorders) | 48 | 37
ASTHENIA (General disorders) | 32 | 31
FATIGUE (General disorders) | 54 | 43
MUCOSAL INFLAMMATION (General disorders) | 22 | 8
PYREXIA (General disorders) | 39 | 30
HYPERSENSITIVITY (Immune system disorders) | 13 | 1
PARONYCHIA (Infections and infestations) | 20 | 0
WEIGHT DECREASED (Investigations) | 26 | 19
ANOREXIA (Metabolism and nutrition disorders) | 34 | 23
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 10 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 11 | 5
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 16 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 | 8
DIZZINESS (Nervous system disorders) | 11 | 3
HEADACHE (Nervous system disorders) | 11 | 8
NEUROPATHY (Nervous system disorders) | 10 | 16
NEUROTOXICITY (Nervous system disorders) | 12 | 7
PARAESTHESIA (Nervous system disorders) | 19 | 38
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 46 | 51
POLYNEUROPATHY (Nervous system disorders) | 9 | 5
INSOMNIA (Psychiatric disorders) | 9 | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 | 7
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 15 | 11
ACNE (Skin and subcutaneous tissue disorders) | 10 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 21 | 17
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 38 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 28 | 3
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 12 | 0
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 11 | 2
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 19 | 7
PRURITUS (Skin and subcutaneous tissue disorders) | 15 | 6
RASH (Skin and subcutaneous tissue disorders) | 90 | 4
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 17 | 0
SKIN TOXICITY (Skin and subcutaneous tissue disorders) | 13 | 0
HYPERTENSION (Vascular disorders) | 11 | 8

LIMITATIONS AND CAVEATS:
A non-specific outcome measure 'Safety' was deleted from this entry in error. A replacement outcome has been created. The 'Safety' outcome refers to adverse events and these are shown in the 'Adverse Events' section.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days